CLINICAL TRIAL: NCT01437033
Title: A Pilot Study of a Breath Test for Assessment of Volatile Organic Compounds
Brief Title: Breath Test for Chemicals (Volatile Organic Compounds)
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911243; 11-C-N243
Record Dates: First submitted 2011-09-16; First posted 2011-09-20 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2016-09-23

CONDITIONS: Breath Tests; Human Volunteers; Pilot Study
Keywords: Breath Tests; Human Volunteers; Pilot Study; Breath Test

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
Background:

- Some types of cancer, like cancer of the esophagus, are difficult to detect at an early stage. A possible detection method involves collecting breath samples to look for chemicals that may be signs of cancer. However, more research is needed to determine how different chemicals appear in different breath samples. This study will involve healthy volunteers.

Objectives:

- To study chemicals appearing in breath samples of healthy volunteers.

Eligibility:

- Healthy volunteers between 30 and 60 years of age.

Design:

* Participants will fast overnight (midnight to morning) and then provide two breath samples taken 5 minutes apart.
* Breath samples will be collected on days 1, 49, and 98 of the study

DETAILED DESCRIPTION:
Background:

Although breath tests are common for specific uses where the biomarker is highly concentrated (e .g. alcohol, urea for Helicobacter prylori infection), lower concentration compounds in the breath can also provide information on exogenous exposures and endogenous metabolic processes.

Employing standardized collection techniques and high sensitivity measurement technologies have shown that breath profiles can accurately identify people with diseases such as breast cancer and lung cancer.

Breath profiling technologies have great potential as non-invasive tools for diagnosis and risk stratification of precancerous disease as well as elucidation of the causes of cancer.

Prior to using breath profiles for these purposes it is essential to assess how much of the breath profile and which parts of the breath profile are relatively stable over a period of time.

Objectives:

The primary objective of this pilot study is to assess the intra-individual variability of breath profiles sampled over a period of 98 days.

Eligibility:

DCEG volunteers aged 30-60 years, inclusive.

Design:

Pilot study.

Five DCEG volunteers will be enrolled for this study.

We will assess breath profiles sampled in duplicate at three time periods (days 1, 49 and 98).

We will calculate a coefficients of variation (CV) to determine the proportion and parts of the breath profile which have values less than 10% when collected on the same day,49 days apart, and 98 days apart.

ELIGIBILITY:
* INCLUSION CRITERIA:

DCEG volunteers aged 30-60 years, inclusive.

EXCLUSION CRITERIA:

Aged less than 30 years. Aged 61 years or older. Individuals who identify themselves to be in any one of the following categories over the next 4 month period:

* Plan to initial a large change in their daily amount of physical activity
* Plan to make large changes to their diet (reduce caloric intake, become a vegetarian etc)
* May possibly move away from the area for a new job, sabbatical, retirement etc
* Plan to attempt to become pregnant
* Have limited availability for any reason including prolonged vacation or business travel

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2011-08-29; Study Completion 2016-09-23

PRIMARY OUTCOMES:
Statistics of robustness (CV, ICCs) | 98 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Cook, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Cook MB, Dawsey SM, Diaw L, Blaser MJ, Perez-Perez GI, Abnet CC, Taylor PR, Albanes D, Virtamo J, Kamangar F. Serum pepsinogens and Helicobacter pylori in relation to the risk of esophageal squamous cell carcinoma in the alpha-tocopherol, beta-carotene cancer prevention study. Cancer Epidemiol Biomarkers Prev. 2010 Aug;19(8):1966-75. doi: 10.1158/1055-9965.EPI-10-0270. Epub 2010 Jul 20. PMID 20647397
- [Background] Vizcaino AP, Moreno V, Lambert R, Parkin DM. Time trends incidence of both major histologic types of esophageal carcinomas in selected countries, 1973-1995. Int J Cancer. 2002 Jun 20;99(6):860-8. doi: 10.1002/ijc.10427. PMID 12115489
- [Background] Perera FP. Cancer: the big questions to address in coming years. Cancer Epidemiol Biomarkers Prev. 2011 Apr;20(4):571-3. doi: 10.1158/1055-9965.EPI-11-0184. No abstract available. PMID 21454418